CLINICAL TRIAL: NCT04968756
Title: Open Label Early Feasibility Study Evaluating the Safety of the SPECTRALIS CENTAURUS Device for Dosimetry of Selective Retina Therapy With Optical Coherence Tomography
Brief Title: Evaluating the Safety of the SPECTRALIS CENTAURUS Device
Acronym: CENTAURUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Bern University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CENTAURUS
Record Dates: First submitted 2021-04-26; First posted 2021-07-20 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Retinal Diseases
Keywords: Retinal Pigment Epithelium
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with the SPECTRALIS CENTAURUS device (Experimental): In Stage 1, two laser pattern will be applied in areas of the retina that require ablative laser photocoagulation.
  In Stage 2, a laser pattern will be applied along and on the outside of the arcades. Furthermore, a treatment pattern will be applied to an area temporal to the fovea affected by intermediary age-related macular degeneration (AMD) and confluent soft drusen.
  Interventions: Device: Selective retina therapy SPECTRALIS CENTAURUS device

INTERVENTIONS:
Device: Selective retina therapy SPECTRALIS CENTAURUS device — Microsecond laser microsurgery by using the SPECTRALIS CENTAURUS device

SUMMARY:
The objective of this clinical trial is to evaluate the safety of the SPECTRALIS CENTAURUS device (HuCE-optoLab, BFH TI, Biel, CH) in a clinical setting on patients with retinal diseases.

DETAILED DESCRIPTION:
Optical microsurgery of the retinal pigment epithelium (RPE) requires reliable real-time dosimetry to prevent unwanted overexposure of the neuroretina. The SPECTRALIS CENTAURUS device implements optical coherence tomography (OCT) to detect intentional elimination of RPE cells caused by a prototype laser for selective retina therapy (SRT).

Within this clinical trial the safety of the SPECTRALIS CENTAURUS device and its ability to detect RPE cell damage towards selective real-time laser microsurgery will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* For Stage 1, any patient aged >18 years with the need for conventional laser retina ablation
* For Stage 2, will be restricted to people aged 50 to <95 years with lesion characteristics that meet the criteria for intermediate AMD

Exclusion Criteria:

* Presence of reticular pseudodrusen
* Any manifestation of late-stage AMD
* Known hypersensitivity or allergy to fluorescein or uncontrolled hypertension
* Concomitant systemic corticosteroid treatment for continuous period longer than 2 weeks
* History of any vitreous haemorrhage within 4 weeks prior to screening or current haemorrhage in the study eye
* Inability to obtain fundus photographs or fluorescein angiogram of sufficient quality
* Photosensitive epilepsy
* Insufficient retinal pigmentation (albinism)
* Corneal opacity / lens opacity
* Women of child-bearing potential
* Contralateral eye is at an advanced stage of disease and has poor visual acuity
* Inability to follow the procedures of the study
* Participation in another study with investigational drug within the 30 days preceding and during the present study - Inability or lack of willingness to commit to return for all clinical visits and complete all study-related procedures

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety SPECTRALIS CENTAURUS - AEs | 26 weeks
  The primary objective of this study is to assess the safety of the SPECTRALIS CENTAURUS device in clinical use by the evaluation of any adverse events (AEs) that may be related to the study device or the study intervention, including device deficiencies (DDs)
  The following potential AEs are evaluated throughout the study regarding the laser treatment:
  * Decrease in visual acuity
  * Choroidal neovascularization at treatment location (laser lesion)
  * Transient increased edema / decreased vision
  * Development or worsening of macular edema
  * Bruch's membrane rupture
  * Retinal and choroidal haemorrhage
  * Inadvertent foveal burns
Safety SPECTRALIS CENTAURUS - DDs | At treatment (baseline)
  In addition to the AEs, the following potential device deficiencies (DDs) can be listed in relation to the treatment and the SPECTRALIS CENTAURUS device:
  * Unintentional laser delivery
  * Unintentional OCT (M-scan) failure during the treatment
  * Unintentional scanning laser ophthalmoscope (SLO) failure during the treatment
  * Unintentional treatment software failure during the treatment
  * Unintentional treatment laser failure during the treatment
  * Basic system failure during the treatment
  Beside the DDs mentioned above, additional sub-criteria are assessed by default in advance to the treatment visit according to an acceptance test protocol (ATP). The ATP establishes the acceptance test framework for the SPECTRALIS CENTAURUS and describes the scope of the work performed and the approach taken to validate that the system performs as required. An acceptance test is carried out on each day on which a patient is to be treated.

SECONDARY OUTCOMES:
Evaluation of OCT for SRT dosimetry | At treatment (baseline)
  During treatment, OCT M-scans are recorded collinear to the treatment laser application. Post-treatment, all lesions are examined by fluorescein angiography (FA) for RPE cell damage. In addition, the OCT-M scan data is examined for fringe washouts (signal washouts) that occur with RPE cell damage. An analysis of these data (RPE cell damage vs. OCT fringe washouts) will reveal whether OCT is suitable for real-time dosimetry of SRT.
Progression of AMD after laser treatment according to best-corrected visual acuity (BCVA) | At treatment (baseline) and after 1, 4, 12 and 26 weeks
  Course of disease monitoring on AMD and confluent soft drusen with BCVA: Visual acuity is assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart (consisting of rows of letters) / LogMAR chart (Logarithm of the Minimum Angle of Resolution), after appropriate refraction. Visual acuity represents the basic and most clinically relevant functional test to evaluate of central visual acuity.
Progression of AMD after laser treatment according to OCT imaging | At treatment (baseline) and after 1, 4, 12 and 26 weeks
  Course of disease monitoring on intermediary AMD and confluent soft drusen with OCT: OCT provides non-invasive morphological assessment of the retinal layers including the RPE and the choroid. It is a commonly used objective method during clinical assessment. OCT allows to identify structural changes such as Bruch's membrane ruptures, choroidal neovascularizations (CNV) with exudative macular edema, photoreceptor damage and drusen evolution. A macular volume OCT scan centered at the fovea will be acquired routinely. Additionally, volume OCT scans across the laser area will be acquired. This allows, for example, that a change in retinal thickness (μm) can be observed in the short term as well as in the long term. No single endpoint is given for this examination. However, experience shows that CNV would be the most likely case which can be expected with this laser treatment.
Progression of AMD after laser treatment according to FA imaging | At treatment (baseline) and after 12 weeks
  Course of disease monitoring on intermediary AMD and confluent soft drusen with FA: Fluorescein is injected intravenously before serial fundus image are taken after excitation of the fluorescein dye. No single endpoint is given for this examination. However, experience shows that CNV and subtle laser scars would be the most likely cases which can be expected with this laser treatment.
Progression of AMD after laser treatment according to color fundus photography (CFP) | At treatment (baseline) and after 1, 4, 12 and 26 weeks
  Course of disease monitoring on intermediary AMD and confluent soft drusen with CFP: CFP will be used to document and monitor pigmentary changes of the fundus and potential formation of scars after laser application. Since it is difficult to quantify fundus image changes, the principal investigator as well as a safety committee will evaluate fundus changes on an individual basis, taking into account the location and laser parameters used in the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Dysli, MD PhD, Principal Investigator — University of Bern
Locations (1):
- University Hospital Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No